CLINICAL TRIAL: NCT02138825
Title: A Randomized, Double-blind, Placebo-controlled Phase II Study to Investigate the Efficacy and Safety of Riociguat (0.5 mg, 1.0 mg, 1.5 mg, 2.0 mg and 2.5 mg TID) in Patients With Symptomatic Pulmonary Hypertension Associated With Idiopathic Interstitial Pneumonias (IIP).
Brief Title: Efficacy and Safety of Riociguat in Patients With Symptomatic Pulmonary Hypertension (PH) Associated With Idiopathic Interstitial Pneumonias (IIP)
Acronym: RISE-IIP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated per recommendation of iDMC. On iDMC request, protocol amended to include 4-month safety follow-up for patients after withdrawal of riociguat.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13605; 2010-024332-42 (EudraCT Number)
Record Dates: First submitted 2014-04-15; First posted 2014-05-15 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-10

CONDITIONS: Idiopathic Interstitial Pneumonias / Hypertension,Pulmonary
MeSH Terms: conditions — Idiopathic Interstitial Pneumonias; Hypertension | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Riociguat (Adempas, BAY63-2521) (Experimental): In the main study treatment phase participants received Riociguat titrated to optimal dose within range of 0.5 mg TID (3 times a day) to 2.5 mg TID for 10 weeks followed by maintenance period of 16 weeks. This phase was followed by a long-term extension phase, which included a blinded sham titration phase of 10 weeks followed by an open-label extension phase. During the open-label extension phase participants were to be treated with Riociguat until commercial access in the indication of pulmonary hypertension (PH) associated with idiopathic interstitial pneumonias (IIP) or until an agreed time point is defined with the individual country, local regulatory authority and the Sponsor's global team.
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)
- Placebo (Placebo Comparator): In the main study treatment phase participants received sham titration within range of 0.5 mg TID to 2.5 mg TID for 10 weeks followed by maintenance period of 16 weeks. This phase was followed by a long-term extension phase, which included a blinded titration phase to optimal dose of Riociguat of 10 weeks followed by an open-label extension phase. During the open-label extension phase participants were to be treated with Riociguat until commercial access in the indication of PH associated with IIP or until an agreed time point is defined with the individual country, local regulatory authority and the Sponsor's global team.
  Interventions: Drug: Riociguat (Adempas, BAY63-2521); Drug: Placebo

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — Active drug 0.5 mg, 1.0 mg, 1.5 mg, 2.0 mg and 2.5 mg TID/day as per individual dose titration. The starting dose will be 0.5 mg TID, and the dose will be adjusted every two weeks for ten weeks in 0.5 mg increments up to a maximum dose of 2.5 mg TID based on patient's systolic blood pressure and well-being.
Drug: Placebo — Inactive dosed at 0.5 mg, 1.0 mg, 1.5 mg, 2.0 mg and 2.5 mg TID/day as per individual dose titration for 26 weeks
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of 26-weeks of treatment with riociguat vs. placebo in patients with symptomatic PH (pulmonary hypertension) associated with IIP (idiopathic interstitial pneumonias).

DETAILED DESCRIPTION:
Number of participants with Adverse Events (AEs) will be reported in Adverse Events section.

ELIGIBILITY:
* Inclusion Criteria:
* Men or women aged from ≥18 to ≤80 years
* Diagnosed with one of the following (confirmed using a multidisciplinary approach, as per ATS(American Thoracic Society) / ERS(European Respiratory Society) / JRS (Japanese Respiratory Society) / ALAT(Latin American Thoracic Association) guidelines:

  * Major IIPs (idiopathic interstitial pneumonias) diagnosis or suspected as one of the following:
  * Idiopathic pulmonary fibrosis
  * Idiopathic nonspecific interstitial pneumonia
  * Respiratory bronchiolitis-interstitial lung disease
  * Desquamative interstitial pneumonia
  * Cryptogenic organizing pneumonia
  * Acute interstitial pneumonia
  * Rare IIPs diagnosis by one of the following:
  * Idiopathic lymphoid interstitial pneumonia
  * Idiopathic pleuroparenchymal fibroelastosis
  * Unclassifiable idiopathic interstitial pneumonias
* Forced Vital Capacity (FVC) ≥ 45 %
* 6MWD (6 minutes walking distance) ≥ 150 m to ≤ 450 m {under stable O2(oxygen) supplementation via nasal cannula}
* Diagnosis of PH (pulmonary hypertension) confirmed by right heart catheter (RHC) with (mean artery pulmonary artery pressure )mPAP ≥ 25 mmHg and (pulmonary artery wedge pressure)PAWP ≤15 mmHg at rest
* Systolic blood pressure (SBP) ≥ 95 mmHg and no signs or symptoms of hypotension
* WHO functional class II-IV
* Women of childbearing potential can only be included in the study if a pregnancy test is negative. Women of childbearing potential must agree to use adequate contraception when sexually active. 'Adequate contraception' is defined as any combination of at least 2 effective methods of birth control, of which at least one is a physical barrier (e.g. condoms with hormonal contraception or implants or combined oral contraceptives, certain intrauterine devices). Adequate contraception is required from the signing of the informed consent form up until 4 weeks after the last study drug administration
* Exclusion Criteria:
* Known significant left heart disease:

  * Pulmonary venous hypertension indicated by baseline pulmonary capillary wedge pressure > 15 mmHg
  * Symptomatic coronary artery disease
  * Systolic left-ventricular dysfunction with an left ventricular ejection fraction (LVEF) <45%
* Active state of hemoptysis or pulmonary hemorrhage, including those events managed by bronchial artery embolization
* Any history of bronchial artery embolization or massive hemoptysis within 3 months prior to screening. Massive hemoptysis being defined as acute bleeding >240 mL in a 24-hour period or recurrent bleeding >100 mL/d over several days
* Difference > 15% between the eligibility and the baseline 6MWD test
* Forced expiratory volume in one second (FEV1) / Forced Vital Capacity (FVC) <0.65 after bronchodilator administration
* Initiation in cytotoxic, immunosuppressive, cytokine modulating therapy initiated within 3 months prior to screening. Such agents might include. azathioprine, cyclophosphamide, corticosteroids, etanercept, tumor necrosis factor alpha (TNFα) inhibitors and others
* Any specific treatment for (pulmonary arterial hypertension) PAH/PH (pulmonary hypertension )within 3 months prior to screening
* Concomitant use of the following medication: nitrates or (nitric oxide) NO donors (such as amyl nitrite) in any form, phosphodiesterase 5 inhibitors (such as sildenafil, tadalafil, vardenafil) and non-specific phosphodiesterase (PDE) inhibitors (theophylline, dipyridamole),
* Pregnant women (i.e. positive pregnancy test or other signs of pregnancy), or breast feeding women, or women of childbearing potential not using adequate contraception (as defined in the aforementioned inclusion criterion) and not willing to agree to 4 weekly pregnancy testing from Visit 1(first administration of study drug) onwards until 4 weeks after last study drug intake

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2014-06-04 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (87):
- United States (17):
  - University of California, Los Angeles, Los Angeles, California
  - San Francisco, California
  - Aurora, Colorado
  - Miami, Florida
  - Orlando, Florida
  - Via Christi Clinic, Wichita, Kansas
  - Louisville, Kentucky
  - Columbia University Medical Center, New York, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Falls Church, Virginia
- Argentina (4):
  - Mar del Plata, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Godoy Cruz, Mendoza Province
  - San Miguel de Tucumán, Tucumán Province
- Australia (7):
  - Camperdown, New South Wales
  - Darlinghurst, New South Wales
  - Sydney, New South Wales
  - Chermside, Queensland
  - Adelaide, South Australia
  - Prahran, Victoria
  - Murdoch, Western Australia
- Leuven, Belgium
- Canada (4):
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Toronto, Ontario
  - Québec
- Colombia (4):
  - Bogotá, Bogota D.C.
  - Floridablanca-Bucaramanga, Santander Department
  - Cali, Valle del Cauca Department
  - Bogotá
- Aarhus N, Denmark
- France (4):
  - Bron
  - Lille
  - Marseille
  - Paris
- Germany (7):
  - München, Bavaria
  - Würzburg, Bavaria
  - Giessen, Hesse
  - Hanover, Lower Saxony
  - Essen, North Rhine-Westphalia
  - Dresden, Saxony
  - Großhansdorf
- Greece (4):
  - Athens
  - Haidari
  - Ioannina
  - Thessaloniki
- Israel (4):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
- Italy (5):
  - Forlì-Cesena, Emilia-Romagna
  - Rome, Lazio
  - Monza-Brianza, Lombardy
  - Palermo, Sicily
  - Siena, Tuscany
- Japan (5):
  - Seto, Aichi-ken
  - Yokohama, Kanagawa
  - Sakai, Osaka
  - Shibuya-ku, Tokyo
  - Chiba
- New Zealand (2):
  - Auckland
  - Christchurch
- Portugal (3):
  - Coimbra
  - Porto
  - Vila Nova de Gaia
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Vladimir
- Riyadh, Saudi Arabia
- Spain (2):
  - Barcelona
  - Valencia
- Switzerland (3):
  - Bern
  - Geneva
  - Zurich
- Turkey (Türkiye) (2):
  - Denizli
  - Izmir
- United Kingdom (4):
  - Cambridge, Cambridgeshire
  - Clydebank, West Dunbartonshire
  - London
  - Newcastle

REFERENCES:
- [Derived] Nathan SD, Behr J, Collard HR, Cottin V, Hoeper MM, Martinez FJ, Corte TJ, Keogh AM, Leuchte H, Mogulkoc N, Ulrich S, Wuyts WA, Yao Z, Boateng F, Wells AU. Riociguat for idiopathic interstitial pneumonia-associated pulmonary hypertension (RISE-IIP): a randomised, placebo-controlled phase 2b study. Lancet Respir Med. 2019 Sep;7(9):780-790. doi: 10.1016/S2213-2600(19)30250-4. Epub 2019 Aug 12. PMID 31416769
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 229 participants were enrolled into the study centers in 19 countries worldwide, from 04-Jun-2014 (first patient first visit) to 14-Sep-2016 (last patient last visit).
Pre-assignment Details: A total of 147 participants were randomized and entered the main study phase, of whom 73 were assigned to riociguat and 74 to placebo.
Groups:
- Riociguat (Adempas, BAY63-2521): In the main study treatment phase participants received Riociguat titrated to optimal dose within range of 0.5 mg TID (3 times a day) to 2.5 mg TID for 10 weeks followed by maintenance period of 16 weeks. This phase was followed by a long-term extension (LTE) phase, which included a blinded sham titration phase of 10 weeks followed by an open-label extension phase. During the open-label extension phase participants were to be treated with Riociguat until commercial access in the indication of pulmonary hypertension (PH) associated with idiopathic interstitial pneumonias (IIP) or until an agreed time point is defined with the individual country, local regulatory authority and the Sponsor's global team.
- Placebo: In the main study treatment phase participants received sham titration within range of 0.5 mg TID to 2.5 mg TID for 10 weeks followed by maintenance period of 16 weeks. This phase was followed by a long-term extension (LTE) phase, which included a blinded titration phase to optimal dose of Riociguat of 10 weeks followed by an open-label extension phase. During the open-label extension phase participants were to be treated with Riociguat until commercial access in the indication of PH associated with IIP or until an agreed time point is defined with the individual country, local regulatory authority and the Sponsor's global team.
Period: Main Study Treatment
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Started | 73 (safety population) | 74 (safety population)
Completed | 33 | 39
Not Completed | 40 | 35
Not completed — Adverse Event | 11 | 3
Not completed — Death | 1 | 2
Not completed — Protocol Violation | 2 | 2
Not completed — Sponsor decision | 12 | 18
Not completed — Study terminated by sponsor | 10 | 9
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Medical decision | 1 | 0
Period: Long-term Extension
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Started | 32 | 38
Completed | 0 (no participants were considered as completed LTE phase at time of study termination) | 0 (no participants were considered as completed LTE phase at time of study termination)
Not Completed | 32 | 38
Not completed — Study termination by sponsor | 32 | 38
Period: Safety Follow-up
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Started | 72 (Participants from main study treatment and LTE phase entered safety follow-up) | 64 (Participants from main study treatment and LTE phase entered safety follow-up)
Completed | 50 | 47
Not Completed | 22 | 17
Not completed — Adverse Event | 4 | 3
Not completed — Death | 11 | 5
Not completed — Withdrawal by Subject | 5 | 3
Not completed — clinic worsening | 1 | 0
Not completed — withdrawal by PI | 1 | 0
Not completed — logistical difficulties | 0 | 1
Not completed — progressive disease | 0 | 2
Not completed — too unwell to attend the visit | 0 | 1
Not completed — treatment unblinded | 0 | 1
Not completed — withdrawn due to lung transplant | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo | Total
Number analyzed (Participants) | 73 | 74 | 147
Age, Customized [Number; unit: Participants]
  <65 years | 20 | 17 | 37
  >=65 - <75 years | 35 | 45 | 80
  >=75 years | 18 | 12 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 29 | 52
  Male | 50 | 45 | 95
Pulmonary hypertension (PH) subtype (Nice Clinical Classification) [Number; unit: Participants]
  PH owing to respiratory disease and /or hypoxia | 73 | 74 | 147
  Other | 0 | 0 | 0
Classification of Idiopathic Interstitial Pneumonia [Number; unit: Participants]
  Idiopathic pulmonary fibrosis | 54 | 49 | 103
  Idiopathic nonspecific interstitial pneumonia | 9 | 14 | 23
  Resp. bronchiolitis-interstitial lung disease | 1 | 0 | 1
  Cryptogenic organizing pneumonia | 0 | 1 | 1
  Acute interstitial pneumonia | 0 | 1 | 1
  Idiopathic lymphoid interstitial pneumonia | 0 | 2 | 2
  Unclassifiable idiopathic interstitial pneumonias | 9 | 7 | 16
World Health Organization (WHO) functional class [Number; unit: Participants] — The WHO functional assessment of pulmonary arterial hypertension ranged from functional class I (Patients with PH but without resulting limitation of physical activity) to class IV (Patients with PH with inability to carry out any physical activity without symptoms. These patients manifest signs of right-heart failure.). Changes to a lower WHO functional class resemble improvement, changes to a higher functional class resemble deterioration of pulmonary arterial hypertension (PAH).
  Participants
    Class II | 16 | 22 | 38
    Class III | 50 | 45 | 95
    Class IV | 7 | 7 | 14
6 minute walking distance (6MWD) category [Number; unit: Participants] — The 6MWD test is designed to evaluate a patient's exercise capacity while performing an everyday activity.
  Participants
    < 320 m | 43 | 32 | 75
    >= 320 m and <380m | 12 | 28 | 40
    >= 380 m | 18 | 14 | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in 6 Minute Walking Distance (6MWD) From Baseline to Week 26
Description: The 6MWD test is designed to evaluate a patient's exercise capacity while performing an everyday activity.
Time Frame: Baseline to 26 weeks
Population: Intent to treat (ITT) analysis set: participants randomized and received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 73 | 74
Meter | 3.63 (60.80) | -15.94 (63.70)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) vs Placebo; The evaluation of primary efficacy endpoint will be based on change from baseline in 6MWD using analysis of covariance (ANCOVA) with baseline 6MWD, treatment arm and region as factors; Test type: Superiority or Other; p = 0.2074, ANCOVA; LS mean difference = 21.48, 95% CI 2-sided [-8.75 to 51.71]

2. Secondary Outcome: Number of Participants With Clinical Worsening
Description: The combined endpoint "time to clinical worsening", made up of the following components, defined by the first occurrence: all-cause mortality; need for hospitalization due to worsening cardiopulmonary (CP) status, attributable to progression of disease (including but not limited to increased shortness of breath or increased leg swelling); >15% decrease in the 6MWD test; worsening of WHO functional class.
Time Frame: From baseline to week 26
Population: Intent to treat (ITT) analysis set: participants randomized and received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 73 | 74
Participants
  No clinical event | 39 | 38
  >15% decrease in 6MWD | 9 | 17
  All-cause mortality | 1 | 0
  Hospitalization due to worsening CP status | 15 | 7
  Worsening of WHO functional class | 9 | 12
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) vs Placebo; The difference in incidences in clinical worsening and mortality will be analyzed using Mantel-Haenszel weights, stratified by region; Test type: Superiority or Other; p = 0.3437, Mantel Haenszel

3. Post Hoc Outcome: Number of Deaths Per Study Phase for Riociguat Group
Description: In the main study treatment phase participants received Riociguat until 26 weeks. This phase was followed by a long-term extension (LTE) phase, during which participants continued with Riociguat treatment. At the time of study termination, all treated participants were taken off study drug and started the safety follow-up phase, regardless of whether they were in the main phase or in the LTE.
Time Frame: From start of treatment to end of study
Population: Intent to treat (ITT) analysis set: participants randomized and received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Riociguat (Adempas, BAY63-2521)
Number analyzed (Participants) | 73
Participants
  Main study treatment | 8
  Long-term extension | 1
  Safety follow-up | 3

4. Post Hoc Outcome: Number of Deaths Per Study Phase for Placebo Group
Description: In the main study treatment phase participants received Placebo until 26 weeks. This phase was followed by a long-term extension (LTE) phase, during which participants were treated with Riociguat. At the time of study termination, all treated participants were taken off study drug and started the safety follow-up phase, regardless of whether they were in the main phase or in the LTE.
Time Frame: From start of treatment to end of study
Population: Intent to treat (ITT) analysis set: participants randomized and received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo
Number analyzed (Participants) | 74
Participants
  Main study treatment | 3
  Long-term extension: received Riociguat | 8
  Safety follow-up: only treated with Placebo | 3
  Safety follow-up: received Riociguat in LTE | 1

5. Post Hoc Outcome: Number of Serious Adverse Events During Safety Follow-up Phase
Description: At the time of study termination, all participants entered safety follow-up phase regardless of whether they were in the main phase or in the LTE. Participants who had the End of Treatment visit prior to the implementation of the 120-day safety follow-up were followed-up for at least 30 days.
Time Frame: From start of safety follow-up phase until end of study
Population: Safety analysis set: participants randomized and received at least one dose of study medication.
Measure: Number; unit: Participants
Groups:
- Riociguat up to 2.5 mg Tid: All participants that were initially randomized to Rioiciguat treatment were taken off study drug at the time of study termination, and started the 120 days safety follow-up phase, regardless of whether they were in the main phase or in the LTE. Participants who had the End of Treatment visit prior to the implementation of the 120-day safety follow-up were followed-up for at least 30 days.
- Placebo: All participants that were initially randomized to placebo were taken off study drug at the time of study termination, and started the 120 days safety follow-up phase, regardless of whether they were in the main phase or in the LTE. Participants who had the End of Treatment visit prior to the implementation of the 120-day safety follow-up were followed-up for at least 30 days.
Arm/Group | Riociguat up to 2.5 mg Tid | Placebo
Number analyzed (Participants) | 73 | 74
Participants | 18 | 14

ADVERSE EVENTS:
Time Frame: Treatment emergent Adverse Events are reported: from start of study treatment up to 7 days after end of treatment.
Description: Participants in Placebo group were transitioned to Riociguat treatment in LTE phase.
Groups:
- Riociguat up to 2.5 mg Tid: Reporting group 1 (RG 1): All participants randomized to Riociguat treatment in Main study treatment phase (data until week 26); participants received Riociguat titrated to optimal dose within range of 0.5 mg TID to 2.5 mg TID for 10 weeks followed by maintenance period of 16 weeks. Note: safety data presented here include participants in Riociguat Arm of Period 1 in Participant Flow section.
- Placebo: Reporting group 2 (RG 2): All participants randomized to Placebo treatment in Main study treatment phase (data until week 26); participants received sham titration within range of 0.5 mg TID to 2.5 mg TID for 10 weeks followed by maintenance period of 16 weeks. Note: safety data presented here include participants in Placebo Arm of Period 1 in Participant Flow section.
- Riociguat-Riociguat Transition: Reporting group 3 (RG 3): All participants that were initially randomized to Riociguat treatment in Main study treatment phase and later entered Long-term extension (LTE) phase (data starting from week 26 to study termination); participants received a blinded sham titration phase of 10 weeks followed by an open-label extension phase. During the open-label extension phase participants were to be treated with Riociguat until the study was terminated. Note: safety data presented here include participants in Riociguat Arm of Period 2 in Participant Flow section.
- Placebo-Riociguat Transition: Reporting group 4 (RG 4): All participants that were initially randomized to Placebo treatment in Main study treatment phase and later entered LTE phase (data starting from week 26 to study termination); participants received a blinded titration phase to optimal dose of Riociguat of 10 weeks followed by an open-label extension phase. During the open-label extension phase participants were to be treated with Riociguat until the study was terminated. Note: safety data presented here include participants in Placebo Arm of Period 2 in Participant Flow section.
Arm/Group | Riociguat up to 2.5 mg Tid | Placebo | Riociguat-Riociguat Transition | Placebo-Riociguat Transition
Serious Adverse Events (participants affected / at risk) | 27/73 | 17/74 | 12/32 | 21/38
Other Adverse Events (participants affected / at risk) | 54/73 | 52/74 | 26/32 | 32/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Riociguat up to 2.5 mg Tid (N=73) | Placebo (N=74) | Riociguat-Riociguat Transition (N=32) | Placebo-Riociguat Transition (N=38)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Nodal rhythm (Cardiac disorders) | 1 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 2 | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Choroidal neovascularisation (Eye disorders) | 0 | 1 | 0 | 0
Neovascular age-related macular degeneration (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Incarcerated hernia (General disorders) | 0 | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1 | 0 | 4
Pneumonia moraxella (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Bone abscess (Infections and infestations) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral artery thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 0 | 0 | 1 | 0
Lung transplant (Surgical and medical procedures) | 2 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Riociguat up to 2.5 mg Tid (N=73) | Placebo (N=74) | Riociguat-Riociguat Transition (N=32) | Placebo-Riociguat Transition (N=38)
Right ventricular failure (Cardiac disorders) | 4 | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 4 | 2 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 11 | 7 | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 1 | 1 | 3
Nausea (Gastrointestinal disorders) | 10 | 9 | 4 | 5
Vomiting (Gastrointestinal disorders) | 8 | 2 | 3 | 4
Chest pain (General disorders) | 4 | 5 | 2 | 1
Fatigue (General disorders) | 3 | 7 | 3 | 2
Oedema peripheral (General disorders) | 15 | 7 | 5 | 5
Bronchitis (Infections and infestations) | 2 | 3 | 2 | 2
Influenza (Infections and infestations) | 0 | 1 | 2 | 3
Lower respiratory tract infection (Infections and infestations) | 4 | 1 | 2 | 2
Nasopharyngitis (Infections and infestations) | 5 | 4 | 1 | 3
Sinusitis (Infections and infestations) | 0 | 2 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 2 | 2 | 0
Respiratory tract infection (Infections and infestations) | 6 | 6 | 1 | 2
Blood glucose increased (Investigations) | 3 | 1 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 3 | 7 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 0
Dizziness (Nervous system disorders) | 7 | 8 | 5 | 5
Headache (Nervous system disorders) | 8 | 9 | 2 | 2
Presyncope (Nervous system disorders) | 2 | 1 | 2 | 1
Syncope (Nervous system disorders) | 3 | 2 | 1 | 4
Insomnia (Psychiatric disorders) | 2 | 1 | 1 | 4
Renal failure (Renal and urinary disorders) | 1 | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 6 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 0
Hypotension (Vascular disorders) | 4 | 1 | 3 | 7
Angina unstable (Cardiac disorders) | 0 | 0 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 2 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 3
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 3
Catheterisation cardiac (Investigations) | 0 | 0 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated following a recommendation from the independent Data Monitoring Committee, as patients receiving Riociguat showed an increased risk of mortality and serious adverse events as compared to patients receiving Placebo

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Written consent must be obtained from Bayer prior to any information being submitted for publication. Material proposed for publication or presentation must be provided to Bayer prior to submission. All reasonable comments made by the Sponsor in relation to a proposed publication by the Investigator will be incorporated by the Investigator into the publication.